CLINICAL TRIAL: NCT06538662
Title: A Multicenter, Randomized, Double-Masked, Vehicle-Controlled, Parallel-Group Efficacy and Safety Study of FID 123320 Ophthalmic Solution for the Reduction of Ocular Redness in Pediatric and Adult Populations
Brief Title: An Investigation of FID 123320 for the Reduction of Ocular Redness in Pediatric and Adult Populations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEW422-C003
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Ocular Redness; Eye Irritation
Keywords: Reduction of ocular redness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- FID 123320 Ophthalmic Solution - Adult Cohort (Experimental): 1 drop instilled in each eye at Visit 2 (Day 1), followed by one drop instilled in each eye twice a day (approximately 12 hours apart) Day 2 up to Visit 5 (Day 56), followed by 1 drop instilled in each eye at Visit 5 (Day 56).
  Interventions: Drug: FID 123320 Ophthalmic Solution
- Vehicle - Adult Cohort (Placebo Comparator): 1 drop instilled in each eye at Visit 2 (Day 1), followed by one drop instilled in each eye twice a day (approximately 12 hours apart) Day 2 up to Visit 5 (Day 56), followed by 1 drop instilled in each eye at Visit 5 (Day 56).
  Interventions: Drug: Vehicle
- FID 123320 Ophthalmic Solution - Pediatric Cohort (Experimental): 1 drop instilled in each eye at Visit 2 (Day 1), followed by one drop instilled in each eye twice a day (approximately 12 hours apart) Day 2 up to Visit 5 (Day 56), followed by 1 drop instilled in each eye at Visit 5 (Day 56).
  Interventions: Drug: FID 123320 Ophthalmic Solution
- Vehicle - Pediatric Cohort (Placebo Comparator): 1 drop instilled in each eye at Visit 2 (Day 1), followed by one drop instilled in each eye twice a day (approximately 12 hours apart) Day 2 up to Visit 5 (Day 56), followed by 1 drop instilled in each eye at Visit 5 (Day 56).
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: FID 123320 Ophthalmic Solution — Investigational sterile aqueous solution
  Arms: FID 123320 Ophthalmic Solution - Adult Cohort; FID 123320 Ophthalmic Solution - Pediatric Cohort
Drug: Vehicle — FID 123320 Ophthalmic Solution inactive ingredients
  Arms: Vehicle - Adult Cohort; Vehicle - Pediatric Cohort

SUMMARY:
The purpose of this study is to assess the safety and efficacy of FID 123320 Ophthalmic Solution compared to Vehicle for relieving redness of the eye due to minor eye irritations in pediatric and adult populations.

DETAILED DESCRIPTION:
This study will enroll 2 cohorts: An adult cohort (Subjects 18 years and older of age from any race and ethnicity) and a pediatric cohort (Subjects 5 - 17 years of age from any race and ethnicity).

The study will consist of 6 scheduled visits for each cohort: Screening and/or Baseline visit (Day -7 to -1, Visit 1), Eligibility verification/Randomization/1st Treatment visit on Day 1 (Visit 2), 2-week follow-up visit on Day 14 (Visit 3), 4-week follow-up visit on Day 28 (Visit 4), 8-week follow-up/Treatment discontinuation visit on Day 56 (Visit 5), and 7-day follow-up after treatment discontinuation/Exit visit on Day 63 (Visit 6). The primary endpoint will be collected at Day 1 (Visit 2).

The expected study duration for each subject is approximately 10 weeks with approximately 8 weeks (56 days) of investigational product (IP) exposure.

ELIGIBILITY:
Key Inclusion Criteria - Adult Cohort:

* Capable of giving signed informed consent;
* Willing and able to follow all instructions and attend all study visits;
* Able to self-administer eye drops in the opinion of the investigator;
* Have a history of vasoconstrictor (redness relief drop) use within the last 6 months, have an interest in using over-the-counter (OTC) vasoconstrictor eye drops for redness relief, or would benefit from the use of redness relief drops in the opinion of the investigator;
* Ocular health within normal limits, including distance best corrected visual acuity of 20/40 or better in each eye as measured using a Snellen chart;
* Stable ocular health (defined as no ocular conditions requiring therapy or surgical intervention) during the study;
* Other protocol-defined inclusion criteria may apply.

Key Inclusion Criteria - Pediatric Cohort:

* All pediatric subjects: Parent or legal guardian signs informed consent;
* Pediatric subject ages 7-17: Sign an assent form;
* Subject and parent/legal guardian/care giver: Willing and able to follow all instructions and attend all study visits;
* Able to self-administer eye drops satisfactorily or have a subject's care provider or parent/legal guardian at home routinely available for this purpose;
* Ocular health within normal limits; best-corrected visual acuity of 20/40 or better in each eye as measured using a Snellen chart;
* Stable ocular health (defined as no ocular conditions requiring therapy or surgical intervention) during the study;
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria - Pediatric and Adult Cohorts

* Known contraindications or sensitivity to the use of any of the investigational drug(s) or their components, or any other medication required by the protocol;
* Ocular surgical intervention within 6 months prior to Visit 1 (Day -7 to Day -1) or during the study;
* History of lid surgery;
* Ocular condition that, in the opinion of the investigator, could affect the subject's safety or study parameters;
* Other protocol-specified exclusion criteria may apply.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in investigator-assessed ocular redness at 15 minutes post-instillation on Day 1 (Visit 2) - Adult Cohort | Day 1 (Visit 2) pre-instillation; Day 1 (Visit 2) at 15 minutes post-instillation
  Ocular redness will be assessed by the investigator using a 0-4 unit ocular hyperemia scale. This is a co-primary endpoint.
Mean change from baseline in investigator-assessed ocular redness at 10 hours (600 minutes) post-instillation on Day 1 (Visit 2) - Adult Cohort | Day 1 (Visit 2) pre-instillation; Day 1 (Visit 2) at 10 hours (600 minutes) post-instillation
  Ocular redness will be assessed by the investigator using a 0-4 unit ocular hyperemia scale. This is a co-primary endpoint.
Mean change from baseline in investigator-assessed ocular redness at 1 hour (60 minutes) post-instillation on Day 1 (Visit 2) - Pediatric Cohort (12-17 years) | Day 1 (Visit 2) pre-instillation; Day 1 (Visit 2) at 1 hour (60 minutes) post-instillation
  Ocular redness will be assessed by the investigator using a 0-4 unit ocular hyperemia scale.

SECONDARY OUTCOMES:
Mean change from baseline in the investigator-assessed ocular redness at 1 minute post-instillation on Day 1 (Visit 2) - Adult Cohort | Day 1 (Visit 2) pre-instillation; Day 1 (Visit 2) at 1 minute post-instillation
  Ocular redness will be assessed by the investigator using a 0-4 unit ocular hyperemia scale.
Mean change from baseline in the investigator-assessed ocular redness at 8 hours (480 minutes) post-instillation on Day 1 (Visit 2) - Adult Cohort | Day 1 (Visit 2) pre-instillation; Day 1 (Visit 2) at 8 hours (480 minutes) post-instillation
  Ocular redness will be assessed by the investigator using a 0-4 unit ocular hyperemia scale.
Mean change from baseline in the investigator-assessed ocular redness at 12 hours (720 minutes) post-instillation on Day 1 (Visit 2) - Adult Cohort | Day 1 (Visit 2) pre-instillation; Day 1 (Visit 2) at 12 hours (720 minutes) post-instillation
  Ocular redness will be assessed by the investigator using a 0-4 unit ocular hyperemia scale.
Mean change from baseline in the investigator-assessed ocular redness at 30 seconds post-instillation on Day 1 (Visit 2) - Adult Cohort | Day 1 (Visit 2) pre-instillation; Day 1 (Visit 2) at 30 seconds post-instillation
  Ocular redness will be assessed by the investigator using a 0-4 unit ocular hyperemia scale.
Mean change from baseline in investigator-assessed ocular redness at 1 minute post-instillation on Day 1 (Visit 2) - Pediatric Cohort | Day 1 (Visit 2) pre-instillation; Day 1 (Visit 2) at 1 minute post-instillation
  Ocular redness will be assessed by the investigator using a 0-4 unit ocular hyperemia scale. This endpoint is pre-specified for pediatric subjects in the age range of 12-17 years.
Mean change from baseline in investigator-assessed ocular redness at 8 hours (480 minutes) post-instillation on Day 1 (Visit 2) - Pediatric Cohort | Day 1 (Visit 2) pre-instillation; Day 1 (Visit 2) at 8 hours (480 minutes) post-instillation
  Ocular redness will be assessed by the investigator using a 0-4 unit ocular hyperemia scale. This endpoint is pre-specified for pediatric subjects in the age range of 12-17 years.
Mean change from baseline in investigator assessed ocular redness at 30 seconds post-instillation on Day 1 (Visit 2) - Pediatric Cohort | Day 1 (Visit 2) pre-instillation; Day 1 (Visit 2) at 30 seconds post-instillation
  Ocular redness will be assessed by the investigator using a 0-4 unit ocular hyperemia scale. This endpoint is pre-specified for pediatric subjects in the age range of 12-17 years.

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, Pharma, Study Director — Alcon Research, LLC
Locations (10):
- United States (10):
  - Canyon City Eyecare, Azusa, California
  - Eye Research Foundation, Newport Beach, California
  - Vision Institute, Colorado Springs, Colorado
  - Butchertown Clinical Trials, Louisville, Kentucky
  - Andover Eye Associates, Andover, Massachusetts
  - NC Eye Associates, OD, PLLC, Apex, North Carolina
  - CORE, Inc., Shelby, North Carolina
  - Total Eye Care PA, Memphis, Tennessee
  - Advancing Vision Research, LLC, Smyrna, Tennessee
  - Alamo Pediatric Eye Center, PLLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No